CLINICAL TRIAL: NCT03173027
Title: The Efficacy of the Traditional Chinese Medicine Fangji Huangqi Pill Combined With Mobic on Active Knee Osteoarthritis: a Study Protocol for a Randomized, Controlled Clinical Trial
Brief Title: The Efficacy of the Traditional Chinese Medicine Fangji Huangqi Pill Combined With Mobic on Active Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cui xuejun (Other)
Responsible Party: Sponsor-Investigator, Cui xuejun, Clinical research base of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FHP
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Fangji Huangqi Pill; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Drug: Fangji Huangqi pill 4g, twice a day, one month, oral Drug: Mobic 7.5mg, once a day, one month, oral participants should administrate both pill and Mobic
  Interventions: Drug: Fangji Huangqi pill or Fangji Huangqi pill placebo
- Placebo group (Placebo Comparator): Drug: Fangji Huangqi pill placebo 4g, twice a day, one month, oral Drug: Mobic 7.5mg, once a day, one month, oral participants should administrate both pill placebo and Mobic
  Interventions: Drug: Fangji Huangqi pill or Fangji Huangqi pill placebo

INTERVENTIONS:
Drug: Fangji Huangqi pill or Fangji Huangqi pill placebo — For the treatment group (Fangji Huangqi pill group), patients will administrate Fangji Huangqi pill (4 g) in 200 milliliter hot water as the instruction and take the solution orally twice a day for 1 month. While patients in the placebo group will take Fangji Huangqi pill placebo as the same way as the Fangji Huangqi pill group. Besides that, both groups will administrate Mobic (7.5 mg once a day) in addition.

SUMMARY:
Knee osteoarthritis (KOA) is known as degenerative joint disease, which is the most common form of arthritis and the leading cause of disability, loss of function and pain worldwide. Effective therapy to manage RA is still lack at present. Fangji Huangqi pill (FHP) is a Chinese medicine which has been widely used in treating KOA in China for hundreds of years to relieve pain, reduce swelling and protect the affected joints from further degeneration. However, no certain evidence to show the effect of FHP for the management of active KOA.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trials (RCT) will be conducted to explore whether the FHP could relieve pain and protect joints. 200 participants suffering from KOA will be enrolled and treated with FHP or placebo for 1 month. The primary outcome measures are the Visual analogue scale (VAS), Western Ontario and McMaster university of orthopedic index (WOMAC), the Lequesne index, and MOS Sleep Scale would be measured from the baseline to 1 month. The second outcome measures would be the six minutes walking test, the Short Form 36-item Health Survey (SF- 36), the X-ray of both knees, and the adverse events from the baseline to 2 weeks, 4 weeks, and 12 weeks' follow-up. In addition, the VAS score, the WOMAC score, the Lequesne index, and AIS Sleep Scale from the baseline to 2 weeks and 12 weeks' follow-up are also the second outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for knee osteoarthritis (American College of Rheumatology criteria)
* Grade 0-3 on the Kellgren-Lawrence grading system
* No serious medical history
* No known drug allergies
* No steroids, glucosamine, chondroitin sulfate, sodium hyaluronate before Fangji Huangqi pill treatment within 1 month

Exclusion Criteria:

* Combined with other disease such as rheumatoid arthritis, lupus arthritis and et. al
* Grade 4 on the Kellgren-Lawrence grading system
* Allergy to study drug
* Participating in other clinical trial
* Unwilling to give informed consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
change of the visual analogue scale (VAS) | at 1 month
change of the Western Ontario and McMaster university of orthopedic index | at 1 month
change of the Lequesne index | at 1 month
change of the 6 minutes walk test | at 1 month

SECONDARY OUTCOMES:
change of the visual analogue scale (VAS) | from baseline to 2 weeks
change of the visual analogue scale (VAS) | from baseline to 12 weeks
change of the Western Ontario and McMaster university of orthopedic index | from baseline to 2 weeks
change of the Western Ontario and McMaster university of orthopedic index | from baseline to 12 weeks
change of the Lequesne index | from baseline to 2 weeks
change of the Lequesne index | from baseline to 12 weeks
change of the 6 minutes walk test | from baseline to 2 weeks
change of the 6 minutes walk test | from baseline to 12 weeks
change score of the Short Form 36-item Health Survey Questionnaire (SF-36) | from baseline to 2 weeks
change score of the Short Form 36-item Health Survey Questionnaire (SF-36) | from baseline to 4 weeks
change score of the Short Form 36-item Health Survey Questionnaire (SF-36) | from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Longhua Hospital, Shanghai University of TCM, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided